CLINICAL TRIAL: NCT02604355
Title: A Multiple-Center, Randomized, Double-Blind, Placebo-Controlled, Single-Ascending Dose and Multiple-Ascending Dose, Adaptive Parallel Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of RO7020322 Following Oral Administration in Healthy Subjects and Chronic Hepatitis B Patients
Brief Title: A Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of RO7020322 Following Oral Administration in Healthy Participants and Chronic Hepatitis B Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Molecule Development was Terminated
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: BP29948
Record Dates: First submitted 2015-11-10; First posted 2015-11-13 (Estimated); Last update posted 2017-05-25 (Actual); Status verified 2017-05

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Healthy Participants (Multiple-Ascending Dosing) (Experimental)
  Interventions: Other: Matching Placebo; Drug: RO7020322
- Healthy Participants (Single-Ascending Dosing) (Experimental)
  Interventions: Other: Matching Placebo; Drug: RO7020322
- Healthy Participants (Study of Food Effect) (Experimental)
  Interventions: Other: Matching Placebo; Drug: RO7020322
- Participants with Chronic Hepatitis B (Proof of mechanism) (Experimental)
  Interventions: Other: Matching Placebo; Drug: RO7020322

INTERVENTIONS:
Other: Matching Placebo — Oral dosing with placebo capsules to match RO7020322.
Drug: RO7020322 — Adaptive oral dosing with RO7020322 capsules, starting at 1 mg daily, with ascending or adjusted dosing based on the results of previous dosing.

SUMMARY:
This is a multiple-center, randomized, double-blind, placebo-controlled, single-ascending dose and multiple-ascending dose, adaptive parallel study to investigate the safety, tolerability, pharmacokinetics and pharmacodynamics of RO7020322 following oral administration in healthy participants and chronic hepatitis B patients.

ELIGIBILITY:
Inclusion Criteria:

Healthy Participants' Inclusion Criteria:

* A Body Mass Index (BMI) between 18 to 30 kg/m^2, inclusive, and a body weight of at least 50 kg
* Males must agree to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agree to refrain from donating sperm during the study
* Women should be of non-childbearing potential
* Able to comply with study restrictions
* Non-smoker (nor tobacco-containing products) for at least 90 days prior to dosing on Day 1 and agreeing not to smoke during the study

Chronic Hepatitis B-Infected Participants' Inclusion Criteria:

* Chronic hepatitis B infection
* A BMI between 18 to 32 kg/m^2, inclusive
* Positive test for HBsAg for more than 6 months prior to randomization
* On entecavir or tenofovir treatment for at least 6 months prior to randomization and remaining on stable treatment during the study
* Liver biopsy, fibroscan® or equivalent test obtained within the past 6 months demonstrating liver disease consistent with chronic hepatitis B (HBV) infection without evidence of bridging fibrosis or cirrhosis
* Males must agree to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agree to refrain from donating sperm during the study
* Women of childbearing potential must agree to remain abstinent (refrain from heterosexual intercourse) or use non-hormonal contraceptive methods that result in a failure rate of < 1% per year during the treatment period and for at least until the end of the follow-up period

Exclusion Criteria:

Healthy Participants' Exclusion Criteria:

* Women who are lactating
* Any suspicion or history of alcohol and/or other substance abuse or dependence in the past 6 months
* Positive urine drug and alcohol screen (barbiturates, benzodiazepines, methadone, amphetamines, methamphetamines, opiates, cocaine, cannabinoids, and alcohol), or positive cotinine test at Day -1
* Positive result on HBV, hepatitis C (HCV), or human immunodeficiency virus (HIV) 1 and 2
* A personal history of unexplained blackouts or faints, or known risk factors for Torsade de Pointes
* Clinically significant abnormalities (as judged by the Investigator) in the physical examination and in the laboratory test results (including hepatic and renal panels, complete blood count, chemistry panel and urinalysis) at screening and on Day -1
* Participation in an investigational drug or device study within 90 days prior to screening or 5 times the half-life of the investigational drug (whichever is longer)
* Donation of blood over 500 mL within three months prior to screening
* Concomitant disease or condition (including allergic reactions against any drug, or multiple allergies) that could interfere with, or treatment of which might interfere with, the conduct of the study, or that would, in the opinion of the Investigator, pose an unacceptable risk to the healthy participant in this study

Chronic Hepatitis B-Infected Participants' Exclusion Criteria:

* Women who are pregnant (positive pregnancy test) or lactating
* History or other evidence of bleeding from esophageal varices
* Decompensated liver disease
* History or other evidence of a medical condition associated with chronic liver disease other than HBV infection
* Documented history or other evidence of metabolic liver disease within one year of randomization
* Positive test for hepatitis A (IgM anti-HAV), hepatitis C, or HIV
* Documented history of infection with hepatitis D virus
* Expected to need systemic antiviral therapy other than that provided by the study at any time during their participation in the study, with the exception of oral therapy for herpes simplex virus (HSV) I or HSV II
* History of immunologically-mediated disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2015-11-28 (Actual); Primary Completion 2016-05-09 (Actual); Study Completion 2016-05-09 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | Up to 8 weeks
Intensity of adverse events | Up to 8 weeks
Number of participants with clinically significant laboratory abnormalities | Up to 8 weeks
Number of participants with clinically significant electrocardiogram (ECG) abnormalities | Up to 8 weeks
Number of participants with clinically significant vital signs abnormalities | Up to 8 weeks

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of RO7020322 | Up to 18 days
Time from dosing to Cmax (Tmax) of RO7020322 | Up to 18 days
Trough plasma concentrations (Ctrough) of RO7020322 | Up to 18 days
Area under the plasma concentration-time curve between time zero (pre-dose) and the time of the last quantifiable concentration (AUClast) of RO7020322 | Up to 18 days
Area under the plasma concentration-time curve between time zero (pre-dose) extrapolated to infinity (AUC0-Inf) of RO7020322 | Up to 18 days
Apparent clearance (CL/F) of RO7020322 | Up to 18 days
Apparent volume (V/F) of RO7020322 | Up to 18 days
Apparent terminal phase half-life (t1/2) of RO7020322 | Up to 18 days
Area under the plasma concentration-time curve (AUC0-t,ss) of RO7020322 at steady state | Up to 18 days
Area under the plasma concentration-time curve (AUC0-t) of RO7020322 on Day 1 | Up to 18 days
Plasma concentration of hepatitis B surface antigen (HBsAg) | Up to 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (4):
- Queen Mary Hospital, Hong Kong, Hong Kong
- New Zealand (2):
  - Auckland Clinical Studies Limited, Grafton
  - Tauranga Hospital, Tauranga
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Taiwan